CLINICAL TRIAL: NCT01187225
Title: Fibrinogen Concentrate to Treat Bleeding in Children Undergoing Cardiac Surgery With Pump: a Randomised Controlled Clinical Trial
Brief Title: Fibrinogen Concentrate In Children After Cardiac Surgery
Acronym: FiCCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0930/09
Record Dates: First submitted 2010-08-17; First posted 2010-08-24 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Surgical Procedures; Blood Coagulation Disorders; Fibrinogen; Cryoprecipitate
Keywords: Cardiac surgical procedures; Fibrinogen; Bleeding; Cryoprecipitate
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrinogen concentrate (Active Comparator)
  Interventions: Drug: Fibrinogen concentrate
- Cryoprecipitate (Active Comparator)
  Interventions: Drug: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen concentrate — In this arm, children (< 18 year-old)undergoing cardiac surgery with pump will receive fibrinogen concentrate (60 mg/Kg) if they present clinically significant bleeding associated to low levels of fibrinogen (< 1g/L) or TEG < 7 mm
  Other Names: Haemocompletan
  Arms: Fibrinogen concentrate
Drug: Cryoprecipitate — In this arm, children (< 18 year-old)undergoing cardiac surgery with pump will receive cryoprecipiate (10 ml/Kg) if they present clinically significant bleeding associated to low levels of fibrinogen (< 1g/L) or TEG < 7 mm
  Arms: Cryoprecipitate

SUMMARY:
The purpose of this study is to evaluate prospectively whether concentrate fibrinogen reduces blood losses, transfusion requirements and occurrence of clinical complications compared to cryoprecipitate in children after cardiac surgery with pump.

DETAILED DESCRIPTION:
Cardiac surgery in children may be associated with excessive perioperative bleeding. Perioperative excessive bleeding is associated with need of transfusion with allogeneic blood products such as red blood cells, fresh frozen plasma, platelet pools, and cryoprecipitate. Furthermore, bleeding may result in re-exploration, which is associated with increased morbidity and mortality.Recent studies have shown that patients and children undergoing cardiac surgery with pump often experience a significant drop in their levels and function of fibrinogen, and it would be in part responsible for the bleeding. In most centre world-wide, it is common practice to treat bleeding in these patients with cryoprecipitate in order to substitute fibrinogen. Fibrinogen concentrate (Haemocomplettan P)may reduce perioperative bleeding, requirements of blood transfusion and clinical outcomes in children undergoing cardiac surgery with pump, compared to cryoprecipitate.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with pump
* Age until 18 years
* Written informed consent
* Clinically important bleeding in intraoperative
* Fibrinogen lower than 1 g/L or TEG < 7 mm

Exclusion Criteria:

* Previous coagulopathy (clinical history or INR > 1.5)
* Low platelet count (lower than 100.000)
* Product allergy
* Urgent procedures
* Active infection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving any allogeneic blood products | From ICU admission until hospital discharge
  Percentage of patients exposed to allogeneic blood products (red blood cells, FFP, platelet concentrate and cryoprecipitate) after ICU admission until hospital discharge.

SECONDARY OUTCOMES:
Length of ICU stay | Up to ICU discharge
  Length of ICU stay - days since arrival at ICU until discharge
Clinical complications - renal failure, respiratory failure,sepsis, myocardial ischemia, stroke | Up to hospital discharge
  Clinical complications since intraoperative until hospital discharge
Mechanical ventilation free-days | Up to ICU discharge
  Number of days without mechanical ventilation during ICU stay
Length of hospital stay | Up to hospital discharge
  Number of days since arrival at ICU until hospital discharge
Vasopressors free-days | Up to ICU discharge
  Number of days without vasopressors during ICU stay
intraoperative transfusion | intraoperative period
  intraoperative requirements of any blood product (red blood cells, FFP, platelet concentrate and cryoprecipitate))
postoperative blood losses | from ICU admission until hospital discharge
  postoperative blood losses determined by the weight of dressings at intraoperative and chest tube drainage 12h and 24h after ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, São Paulo, Brazil